CLINICAL TRIAL: NCT06888193
Title: A Multicenter Open-label, Prospective Study to Assess the Concentration of Bimekizumab in Mature Breast Milk From Mothers Receiving Treatment With Bimzelx® (Bimekizumab)
Brief Title: A Study to Assess the Concentration of Bimekizumab in Mature Breast Milk From Mothers Receiving Treatment With Bimzelx® (Bimekizumab)
Acronym: BE CARING
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UP0122; 2024-518689-29 (Registry Identifier: EU Clinical Trials); U1111-1318-5063 (Other: World Health Organization (WHO))
Record Dates: First submitted 2025-03-15; First posted 2025-03-21 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Moderate to Severe Plaque Psoriasis; Psoriatic Arthritis; Axial Spondyloarthritis; Hidradenitis Suppurativa
Keywords: Bimekizumab; Breastfeeding mothers; Bimzelx®; PSO; HS; AxSpa; PsA
MeSH Terms: conditions — Arthritis, Psoriatic; Axial Spondyloarthritis; Hidradenitis Suppurativa | interventions — bimekizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bimekizumab (Experimental): Breastfeeding mothers who are already receiving commercial bimekizumab per locally approved prescribing information and in consultation and agreement with their treating physicians will participate in this study. Study participants will continue receiving commercially available bimekizumab under the care of their treating physician.
  Interventions: Drug: Bimekizumab

INTERVENTIONS:
Drug: Bimekizumab — Bimekizumab under the care of their treating physician.
  Other Names: Bimzelx®

SUMMARY:
Primary purpose of the study is to assess the concentration of bimekizumab in mature human breast milk.

ELIGIBILITY:
Inclusion Criteria:

* Study participant must be at least 18 years of age at the time of signing the informed consent.
* Study participant is being treated with commercial bimekizumab per locally approved prescribing information and in accordance with her treating physician.
* Study participant is breastfeeding and intends to breastfeed throughout the Sampling Period.
* The decision to treat with bimekizumab and to breastfeed is made independently from and prior to the study participant consenting to participate in the study.
* Study participant must be on bimekizumab treatment for at least 12 weeks after delivery and since starting/restarting/continuing bimekizumab prior to sampling (prior to start of the Sampling Period).
* A female study participant is eligible to participate if she is not pregnant and does not plan to become pregnant during the study.

Exclusion Criteria:

* Study participant has any medical, obstetrical, or psychiatric condition that, in the opinion of the Investigator, could jeopardize or would compromise the study participant's ability to participate in this study.
* The infant has any abnormality noted on physical examination or medical history that, in the opinion of the Investigator, may jeopardize or compromise study participation.
* Study participant has a history of chronic alcohol or drug abuse within the previous last year.
* Study participant has history of breast implants, breast augmentation, or breast reduction surgery.
* Study participant plans a surgical intervention during the Screening Period and Sampling Period or anticipates having surgery while participating in the Sampling Period (does not apply to tubal ligation).
* Study participant or her infant has participated in another study of an investigational medicinal product (IMP) (and/or an investigational device) within the previous 6 months or is currently participating in another study of an IMP (and/or an investigational device), unless the study is UCB PS0036 or a bimekizumab registry study.
* Study participant or her infant has previously participated (ie, entered the sampling period) in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2027-05-03 (Estimated); Study Completion 2027-05-03 (Estimated)

PRIMARY OUTCOMES:
Concentration of bimekizumab in the breast milk on Day 1 | Day 1
  Breast milk samples will be collected predose on Day 1.
Concentration of bimekizumab in the breast milk on Day 2 | Day 2
  Breast milk samples will be collected predose on Day 2.
Concentration of bimekizumab in the breast milk on Day 3 | Day 3
  Breast milk samples will be collected predose on Day 3.
Concentration of bimekizumab in the breast milk on Day 5 | Day 5
  Breast milk samples will be collected predose on Day 5.
Concentration of bimekizumab in the breast milk on Day 7 | Day 7
  Breast milk samples will be collected predose on Day 7.
Concentration of bimekizumab in the breast milk on Day 9 | Day 9
  Breast milk samples will be collected predose on Day 9.
Concentration of bimekizumab in the breast milk on Day 11 | Day 11
  Breast milk samples will be collected predose on Day 11.
Concentration of bimekizumab in the breast milk on Day 13 | Day 13
  Breast milk samples will be collected predose on Day 13.
Concentration of bimekizumab in the breast milk on Day 15 | Day 15
  Breast milk samples will be collected predose on Day 15.
Concentration of bimekizumab in the breast milk on Day 29 | Day 29
  Breast milk samples will be collected predose on Day 29 for mothers on every 4 weeks (Q4W) dosing regimen.
Concentration of bimekizumab in the breast milk on Day 57 | Day 57
  Breast milk samples will be collected predose on Day 57 for mothers on every 8 weeks (Q8W) dosing regimen.

SECONDARY OUTCOMES:
Estimated Infant Dosage of bimekizumab from breast milk | Predose on Day 1, 2, 3, 5, 7, 9, 11, 13, 15, 29 and 57
  Breast milk samples will be collected predose on Day 1 (bimekizumab dosing day), Days 2, 3, 5, 7, 9, 11, 13, and 15 for all study participants (Day 15 predose if every 2 weeks (Q2W) dosing regimen), predose on Day 29 (if Q4W dosing regimen) or Day 57 (if Q8W dosing regimen).
Relative Infant Dose of bimekizumab from breast milk | Predose on Day 1, 2, 3, 5, 7, 9, 11, 13, 15, 29 and 57
  Breast milk samples will be collected predose on Day 1 (bimekizumab dosing day), Days 2, 3, 5, 7, 9, 11, 13, and 15 for all study participants (Day 15 predose if every 2 weeks (Q2W) dosing regimen), predose on Day 29 (if Q4W dosing regimen) or Day 57 (if Q8W dosing regimen).
Treatment-emergent Adverse Events (TEAEs) of the mother from time of informed consent through SFU contact | From time of informed consent up to approximately 17 weeks
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study medication, whether or not considered related to the study medication.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (10):
- United States (3):
  - Up0122 105, Santa Monica, California
  - Up0122 103, South Miami, Florida
  - Up0122 102, Durham, North Carolina
- Canada (2):
  - Up0122 202, Calgary
  - Up0122 201, Vancouver
- Up0122 303, Herne, Germany
- Spain (2):
  - Up0122 501, Barcelona
  - Up0122 502, Barcelona
- Switzerland (2):
  - Up0122 602, Lausanne
  - Up0122 601, Sankt Gallen

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, individual patient-level data cannot be adequately anonymized as there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.